CLINICAL TRIAL: NCT00518245
Title: A Prospective, Open Label, Randomized, Parallel-group Investigation to Evaluate the Efficacy and Safety of Enoxaparin Versus no Enoxaparin in Subjects With Chest Pain Syndrome and no ECG or Biomarker Abnormalities
Brief Title: Ischemia Driven Enoxaparin Therapy in ACS Presenting as Low Risk (IDEAL)
Acronym: IDEAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low rate of patient recruitment. Cannot achieve sample size.
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr. Anatoly Langer, Chair, Canadian Heart Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRC-022
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Unstable Angina
Keywords: unstable angina; drug therapy; myocardial ischemia; myocardial infarction; hemorrhage
MeSH Terms: conditions — Angina, Unstable; Myocardial Ischemia; Myocardial Infarction; Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: enoxaparin
- 2 (No Intervention)

INTERVENTIONS:
Drug: enoxaparin — Enoxaparin will be given subcutanteously at a dose of 1mg/kg every 12 hours for a minimum of 48 hours (4 doses) and a maximum of 8 days until a diagnostic / therapeutic procedure is performed, or at the discretion of the investigator.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether enoxaparin (an anticoagulant) is effective in the treatment of patients presenting to the emergency room with chest pain and no electrocardiogram or bloodwork evidence of a heart attack, but with other high risk clinical features

DETAILED DESCRIPTION:
Patients with chest pain and abnormal electrocardiogram or bloodwork (biomarker) indicative of a heart attack benefit from anticoagulant therapy such as enoxaparin. However, even patients without abnormalities on the electrocardiogram or bloodwork are at increased risk for heart attack or death, if they have certain clinical risk factors. It is currently not known whether enoxaparin is also beneficial for these patients.

Comparison: enoxaparin in addition to optimal standard care at the discretion of the treating physician, versus optimal standard care without enoxaparin

ELIGIBILITY:
Inclusion Criteria:

* Male or female (negative pregnancy test required for females of childbearing potential) ≥ 18 years of age and capable of signing informed consent;
* Typical chest discomfort at rest; lasting at least 5 minutes in the prior 24 hours that is highly suggestive of myocardial ischemia and is not explained by trauma or obvious abnormalities on chest x-ray;
* Two or more of high-risk clinical features.

Exclusion Criteria:

* Clear indication for low molecular weight or unfractionated heparin;
* Pregnancy;
* Increased bleeding risk;
* Impaired hemostasis;
* Angina from a secondary cause;
* Inability to commence ST segment monitoring within 4 hours of study drug initiation;
* Uninterpretable ST segment based upon baseline 12-lead ECG;
* Any contraindications to treatment with LMWH (or unfractionated heparin), including heparin induced thrombocytopenia, known allergy to heparin, low molecular weight heparin, pork or pork products;
* Renal insufficiency or renal dialysis;
* A prosthetic heart valve;
* Any other clinically relevant serious diseases;
* Current evidence of inebriation with alcohol or intoxication resulting from other drug abuse;
* Treatment with other investigational agents or devices within the previous 30 days, planned use of investigational drugs or devices, or has previously enrolled in this trial;
* Inability to comply with the protocol;
* Inability to understand the nature, scope, and possible consequences of the study or is otherwise unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The incidence of, and time to, the composite endpoint of death, nonfatal MI, recurrent myocardial ischemia, or need for coronary revascularization | 30 days

SECONDARY OUTCOMES:
The incidence of, and time to, the composite endpoint of death, nonfatal MI, recurrent myocardial ischemia, or need for coronary revascularization | 6 months
The incidence of myocardial necrosis (as detected by elevated cardiac troponin I or T). | 24 hours
The incidence of major (including non-CABG-related) and minor hemorrhage. | 48 hours and 30 days
The incidence of all-cause mortality, nonfatal MI, and the combination. | 30 and 180 days
One or more of the followings: hemodynamic instability, congestive heart failure, Clinical need for antithrombotic/antiplatelet therapy beyond aspirin, identifiable culprit lesion on diagnostic coronary angiography | during index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Goodman, MD, MSc, Study Chair — Canadian Heart Research Centre; David Fitchett, MD, Principal Investigator — Unity Health Toronto; Anatoly Langer, MD, MSc, Study Director — Canadian Heart Research Centre; Andrew T Yan, MD, Principal Investigator — Canadian Heart Research Centre
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
insufficient data